CLINICAL TRIAL: NCT00917254
Title: Phase II/III Study of YM150 - A Placebo-controlled, Double-blind, Group Comparison Study in Patients Undergoing Elective Total Knee Replacement Surgery -
Brief Title: Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Knee Replacement Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 150-CL-031
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Venous Thromboembolism
Keywords: YM150; Thrombosis; VTE; Knee Replacement; Anticoagulant; FXa inhibitor
MeSH Terms: conditions — Venous Thromboembolism; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- YM150 group-1 (Experimental): YM150 low dose group
  Interventions: Drug: YM150
- YM150 group-2 (Experimental): YM150 high dose group
  Interventions: Drug: YM150
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- Enoxaparin group (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: YM150 — oral
  Arms: YM150 group-1; YM150 group-2
Drug: Placebo — oral
  Arms: Placebo group
Drug: Enoxaparin — injection
  Arms: Enoxaparin group

SUMMARY:
The purpose of this study is to examine the superiority of YM150 to the placebo and to evaluate the dose-dependent response of YM150 in patients undergoing elective total knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects is scheduled for elective primary total knee replacement surgery
* Written informed consent obtained before screening

Exclusion Criteria:

* Subject has history of deep vein thrombosis and/or pulmonary embolism
* Subject has a hemorrhagic disorder and/or coagulation disorder
* Subject has had clinically important bleeding occurred within 90 days prior to the screening visit
* Subject has an acute bacterial endocarditis, retinopathy, hypertension, or thrombocytopenia
* Subject is receiving anticoagulants/antiplatelets

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Overall incidence of venous thromboembolism | 2 weeks

SECONDARY OUTCOMES:
Incidence of individual venous thromboembolism | 2 weeks
Incidence of bleeding events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (13):
- Japan (7):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu
  - Tōhoku
- Taiwan (4):
  - Changhua
  - Chiayi City
  - Kaohsiung City
  - Taichung
- Thailand (2):
  - Bangkok
  - Chiang Mai